CLINICAL TRIAL: NCT02067403
Title: A Diaphragmatic Electrical Activity Based Optimization Strategy During Pressure Support Ventilation. Effects on Work of Breathing, Patient-ventilator Synchrony and Comparison With Neurally Adjusted Ventilatory Assist
Brief Title: A Diaphragmatic Electrical Activity Based Optimization Strategy During Pressure Support Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB 13-363
Record Dates: First submitted 2014-02-07; First posted 2014-02-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Respiratory Insufficiency
Keywords: Pressure-support; Asynchrony
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eadi optimized pressure-support (Experimental)
  Interventions: Other: Pressure-support Eadi optimization

INTERVENTIONS:
Other: Pressure-support Eadi optimization

SUMMARY:
Pressure support (PS) is a commonly used mode of ventilation which is triggered based upon the patient's own inspiratory efforts. For the most part, pressure support is well tolerated by patients. However, because the trigger for pressure support is an inspiratory effort by the patient, and because the resulting support is constant, the ventilator response can be "out of sync" with the patient's needs. The problem of patient-ventilator asynchrony has been documented to be large in approximately one quarter of patients who require mechanical ventilation. Asynchrony is associated with increased or abnormal work of breathing (WOB) and prolonged duration of mechanical ventilation. Diagnosing asynchrony at the bedside can be challenging. Electrical activation of the diaphragm (Eadi) recording can provide clinicians with a more accurate picture of patient-ventilator synchrony and may thus result in decreased asynchrony and decreased or normalized work of breathing for the patient. The purpose of this physiologic study is to evaluate the role of protocolized pressure support ventilation (based upon Eadi) in comparison to standard pressure support ventilation.

DETAILED DESCRIPTION:
Pressure support will be readjusted according to Eadi recording in different steps.

The optimized pressure support will be compared to the initial pressure support.

ELIGIBILITY:
Inclusion Criteria:

Patients who are ventilated using a partial ventilator support mode (i.e. pressure support) and meet one of the following criteria:

* Known chronic pulmonary obstructive disease
* Suspected Intrinsic PEEP on the expiratory airway pressure and flow tracings
* Resistive pressure (i.e. eak pressure-Plateau pressure) higher than 20 centimeters of water (cmH2O) at a flow of 60 L/min or higher than 15 at a flow of 45 L/min in volume controlled ventilation (preferably after a tracheal aspiration maneuver)
* Known chronic restrictive pulmonary disease with respiratory failure
* Restrictive pulmonary disease characterized by a measured compliance of less than 30 ml/cmH2O
* Obesity with BMI ≥ 30 kg/m2
* Existence of frequent asynchronies noticed on the ventilator waveforms
* Expected duration of ventilation of more than 24 hours

Exclusion Criteria:

* Contraindication to Naso/orogastric tube (NGT/OGT) placement (known esophageal problem such as hiatal hernia or esophageal varicosities, active upper gastro-intestinal bleeding, any other contraindication to the insertion of a NGT/OGT)
* Poor short term prognosis (defined by the clinician in charge as a high risk of death during the next 7 days) or ongoing palliative treatment.
* Patients with "Do not resuscitate" order already established and in palliative care
* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Synchrony and patient effort determined from pressure time product measured from the esophageal pressure | For each step of the protocol (10 minutes/step)

SECONDARY OUTCOMES:
WOB determinated from esophageal pressure measurement using the Campbell diagram | For each step of the protocol (10 minutes/step)
Number of asynchronies | For each step of the protocol (10 minutes/step)
Comfort score (verbal scale) | For each step of the protocol (10 minutes/step)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Beloncle F, Piquilloud L, Rittayamai N, Sinderby C, Roze H, Brochard L. A diaphragmatic electrical activity-based optimization strategy during pressure support ventilation improves synchronization but does not impact work of breathing. Crit Care. 2017 Jan 31;21(1):21. doi: 10.1186/s13054-017-1599-z. PMID 28137269